CLINICAL TRIAL: NCT04773145
Title: Osseointegration of Hydroxyapatite-coated Femoral Stems in Femoral Neck Fractures Over 80 Years
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, Didier MAINARD, Professor, Central Hospital, Nancy, France
Other Study IDs: 2020PI257
Record Dates: First submitted 2021-02-24; First posted 2021-02-26 (Actual); Last update posted 2021-02-26 (Actual); Status verified 2021-02

CONDITIONS: Femoral Neck Fractures
MeSH Terms: conditions — Femoral Neck Fractures | interventions — Hemiarthroplasty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Femoral neck fracture: Patients over 80 years when suffering of femoral neck fracture with at least one year follow-up.
  Interventions: Procedure: Hemiarthroplasty with hydroaxyapatite coated stem

INTERVENTIONS:
Procedure: Hemiarthroplasty with hydroaxyapatite coated stem — Hemiarthroplasty with non cemented femoral stem, using the hydroxyapatite-coated femoral stem Pharo

SUMMARY:
This study aimes to prove that osseointegration of hydroxyapatite coated stem is possible for patients over 80 years with femoral neck fracture, without the risks of cemented stems.

The hydroxyapatite has a local effect which can improve cortical index.

ELIGIBILITY:
Inclusion Criteria:

* 80 years
* 1 year follow-up
* femoral neck fracture

Exclusion Criteria:

* bad-realized radiographs

Min Age: 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: All patients over 80 with femoral neck fracture
Sampling Method: Non-Probability Sample
Enrollment: 140 (Estimated)
Dates: Start 2021-02-24 (Actual); Primary Completion 2021-03-24 (Estimated); Study Completion 2021-03-24 (Estimated)

PRIMARY OUTCOMES:
Engh and Massin score | 1 month
  Measure of the osseointegration

SECONDARY OUTCOMES:
CBR | 1 month
  Mesure of level of osteoporosis

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Hôpital Central, Nancy, Lorraine, France

IPD SHARING:
Plan to Share IPD: Undecided